CLINICAL TRIAL: NCT02503670
Title: HealthyDads.Ca-Development and Pilot Evaluation of a Multimodal E-Health Intervention to Promote the Mental Health of Men at Risk for Depression
Brief Title: An Intervention Study to Evaluate a Website Tailored to New Dads to Promote Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University (Other)
Collaborators: Movember Foundation (Other)
Responsible Party: Principal Investigator, Deborah Da Costa, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Movember A03-B15-14B
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Mental Health in Expectant First-time Fathers
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HealthyDads.ca web-based program (Other): An on-line self-help psychoeducational website tailored to new dads. Psychoeducational learning modules and tools, including a 6 week physical activity challenge..
  Interventions: Behavioral: Psychoeducational modules to prevent/reduce depression
- Control group (Other): No access to the intervention. Will complete the same questionnaires as the Healthydads.ca group over the study period.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Psychoeducational modules to prevent/reduce depression — Psychoeducational learning modules and tools. Men will choose modules based on interest and need.
  Arms: HealthyDads.ca web-based program
Other: Control Group — Continue with standard care.
  Arms: Control group

SUMMARY:
The purpose of this study is to develop and pilot test HealthyDads.ca, a website for expectant first-time fathers who have known risk factors for depression.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate in French or English
* Either married or cohabiting at the time of study entry
* First child for both partners
* Have internet access
* Score <12 on the Edinburgh Postnatal Depression Scale (EPDS)
* Not currently receiving psychotherapy from a health professional or on medication for a mental disorder
* At least 1 risk factor for depression if they score < 6 on the EPDS: a)history of depression, b) elevated anxiety or c) couple discord

Exclusion Criteria:

* Suicidal ideation or intent
* Physical condition precluding participation in exercise

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-12; Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of HealthyDads.caHealthyDads.ca measured by the Usability and Satisfaction questionnaire | 6 weeks post randomization
  To evaluate the acceptability of the internet delivered program in terms of rating on items pertaining to the website's ease of use and satisfaction.
Change from baseline on depressed mood as measured by the Edinburgh Postnatal Depression Scale (EPDS) | Study entry, 6 weeks post randomization, 2 and 6 months following delivery
  This is a widely used reliable and standardized measure of depression.

SECONDARY OUTCOMES:
Changes from baseline on emotional well-being as measured by the Mental Health Continuum-Short Form (MHC-SF) | Study entry, 6 weeks post randomization, 2 and 6 months following delivery
  This is a widely used reliable and standardized measure of psychological well-being.
Changes from baseline on parenting stress measured by the Parenting Stress Scale (PARSS) | Study entry, 6 weeks post randomization, 2 and 6 months following delivery
  This is a widely used reliable and standardized measure of parenting stress.
Changes from baseline on level of physical activity participation measured by the International Physical Activity Questionnaire (IPAQ) | Study entry, 6 weeks post randomization, 2 and 6 months following delivery
  This is a widely used reliable and standardized measure of physical activity.
Changes from baseline on sleep quality measured by the Pittsburgh Sleep Quality Index (PSQI) | Study entry, 6 weeks post randomization, 2 and 6 months following delivery
  This is a widely used reliable and standardized of sleep quality.
Changes from baseline on perceptions of stigma measured with the Stigma Scale for Receiving Psychological Help (SSRPH), | Study entry, 6 weeks post randomization, 2 and 6 months following delivery
  This is a reliable and standardized measure of stigma perceptions associated with with seeking help for mental health issues.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - University of Toronto, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec